CLINICAL TRIAL: NCT02659176
Title: Comparative Study Between Trans-perineal Repair With or Without Limited Internal Sphincterotomy in Treatment of Type I Anterior Rectocele: A Randomized Controlled Trial
Brief Title: Trans-perineal Repair With or Without Limited Internal Sphincterotomy for Treatment of Type I Anterior Rectocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mansoura31
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Rectocele
MeSH Terms: conditions — Rectocele | interventions — CDP-Diacylglycerol-Inositol 3-Phosphatidyltransferase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transperineal repair with PIS (Active Comparator): transperineal repair of anterior rectocele with limited internal sphincterotomy
  Interventions: Procedure: Transperineal repair with PIS
- Transperineal repair without PIS (Active Comparator): transperineal repair of anterior rectocele only
  Interventions: Procedure: Transperineal repair without PIS

INTERVENTIONS:
Procedure: Transperineal repair with PIS — Repair of anterior rectocele via transperineal approach followed by limited internal sphincterotomy at 6 o'clock.
  Arms: Transperineal repair with PIS
Procedure: Transperineal repair without PIS — Repair of anterior rectocele via transperineal approach without performing limited internal sphincterotomy
  Arms: Transperineal repair without PIS

SUMMARY:
Comparison between transperineal repair of rectocele with or without posterior internal sphincterotomy.

DETAILED DESCRIPTION:
Transperineal repair of anterior rectocele is performed in two groups of patients, the first will undergo limited posterior internal sphincterotomy, the second group will not have internal sphincteroromy. The two groups are compared regarding recurrence of rectocele and improvement of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior rectocele

Exclusion Criteria:

* Pregnant females
* Rectocele with pelvic organ prolapse
* Any patient with previous anorectal surgery
* Pudendal nerve neuropathy
* Anal fistula and sepsis
* Patients with sphincter defect proved by endo-anal sonography
* Patients proved to have colonic inertia either by colon transit time and/or history
* Patients with defecography anomalies causing obstructed defecation other than rectocele (e.g. Anismus).
* Also patients with vascular diseases, scleroderma, malnutrition, and coagulopathy were excluded.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrence | 18 months
  Number of patients presenting with recurrent or persistent symptoms during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Youssef, M.D, Principal Investigator — Mansoura Univesity
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No